CLINICAL TRIAL: NCT05361421
Title: Effect of Intensive LDL-cholesterol Targeting for Elderly Patients With Cardiovascular Disease: I-OLD Trial
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 4-2022-0259
Record Dates: First submitted 2022-04-29; First posted 2022-05-04 (Actual); Last update posted 2024-03-15 (Actual); Status verified 2024-03

CONDITIONS: Cardiovascular Disease
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intensive targeting group (Experimental): Intensive lipid loweroing therapy with LDL-cholesterol goal of <55mg/dL
  Interventions: Drug: Intensive targeting group
- Conventional therapy group (Active Comparator): Initiate and maintain moderate intensity statin therapy
  Interventions: Drug: Conventional therapy group

INTERVENTIONS:
Drug: Intensive targeting group — Intensive lipid lowering therapy with LDL-cholesterol goal of <55mg/dL. Atorvastatin 5, 10, 20, 40, and 80mg are allowed to use and ezetimibe or PCSK-9 inhibitor may be considered in patients who could not achieve target LDL-cholesterol level even with the maximum dose of study drugs (atorvastatin 80mg) by the discretion of the investigator.
  Arms: Intensive targeting group
Drug: Conventional therapy group — Only moderate intensity statin therapy (atorvastatin 5, 10, and 20mg ) are allowed. Ezetimibe or PCSK-9 inhibitor is not allowed to use.
  Arms: Conventional therapy group

SUMMARY:
Although there have been studies regarding intensive lowering of low-density lipoprotein (LDL)-cholesterol with high intensity statins in patients with cardiovascular disease, elderly patients were either excluded or accounted only a small portion of study subjects. Therefore, this study sought to compare the clinical outcomes according to the LDL-cholesterol therapy targeting (intensive targeting [LDL-cholesterol <55mg/dL] vs. conventional therapy [moderate intensity statin therapy]) in elderly patients with ≥75 years and documented cardiovascular disease.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥75 years
2. Documented cardiovascular disease (at least 1 of the following) A. Previous acute coronary syndrome (MI or unstable angina) B. Or stable angina with imaging studies of coronary artery disease or functional studies of myocardial ischemia C. Or coronary revascularization (percutaneous coronary intervention or coronary artery bypass graft) D. Or peripheral artery disease.

Exclusion Criteria:

1. MI or stroke within 1 year
2. LDL-cholesterol level less than 55 mg/dL without statin therapy
3. Active liver disease or persistent unexplained serum AST/ALT elevation more than 2 times the upper limit of normal range
4. Allergy or hypersensitivity to any statin
5. Life expectancy less than 1 years
6. Inability to follow the patient over the period of 1 year after enrollment, as assessed by the investigator

Min Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 1200 (Estimated)
Dates: Start 2022-07-19 (Actual); Primary Completion 2025-10-15 (Estimated); Study Completion 2027-10-15 (Estimated)

PRIMARY OUTCOMES:
Clinical efficacy of intensive lipid-lowering therapy | 3 years
  Composite of cardiovascular death, non-fatal myocardial infarction (MI), non-fatal stroke, coronary revascularization, and hospitalization for angina

SECONDARY OUTCOMES:
Efficacy endpoint | 3 years
  1. Each component of primary endpoint
  2. Various composite outcomes A. Composite of cardiovascular death, non-fatal MI, and non-fatal stroke B. Composite of cardiovascular death, non-fatal MI, non-fatal stroke, and coronary revascularization C. Composite of cardiovascular death, non-fatal MI, and coronary revascularization D. Composite of all-cause death, non-fatal MI, non-fatal stroke, coronary revascularization, and hospitalization for angina
  3. Rate of cross-over into the non-allocated therapy regimen (1, 2, and 3 years after enrollment)
Safety endpoint | 3 years
  1. New-onset diabetes mellitus, worsening of glycemic control, or homeostatic model assessment (HOMA)-index
  2. Occurrence of statin-associated muscle symptoms (SAMS) requiring change of therapy regimen or dosage
  3. Elevation of muscle enzymes (CPK > 4 x UNL)
  4. Elevation of hepatic enzymes (AST, ALT, or both ≥ 3 x UNL)
  5. Elevation of serum creatinine level (>50% from baseline)
  6. Change of proteinuria
  7. Diagnosis of cancer
  8. Operation due to cataract
  9. Major bleeding (BARC 2, 3, or 5)

CONTACTS AND LOCATIONS:
Locations (1):
- Yonsei University Health System, Severance Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided